CLINICAL TRIAL: NCT07260045
Title: The Effects of Chiropractic on Adults With Depression: a Pilot Study
Brief Title: The Effects of Chiropractic on Adults With Depression
Acronym: DEP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Life University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: I-0035
Record Dates: First submitted 2025-10-09; First posted 2025-12-02 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-11

CONDITIONS: Depression Disorder
Keywords: Depression; Waitlist; Chiropractic Care
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Waitlist Group (WL) (Other): After the 6-week lab assessments, the participants in the waitlist (WL) group will be offered 6 weeks of chiropractic care.
  Interventions: Other: Chiropractic Care
- Intervention Group (Experimental): Within the 6-week lab assessments, the participants in the intervention group will receive 6 weeks of chiropractic care.
  Interventions: Other: Chiropractic Care

INTERVENTIONS:
Other: Chiropractic Care — Participants of the treatment group will be randomly assigned to chiropractic care for 6 weeks. Participants will have their upper cervical spine (C1/C2) assessed for the presence of vertebral subluxations per the chiropractor's normal and customary procedures.

SUMMARY:
The goal of this clinical trial is to evaluate the feasibility of the study design in preparation for a future clinical trial examining chiropractic care for adults with mild to moderate depression. We aim to determine whether the study procedures function as intended, including the ability to recruit, retain, and engage participants, as well as whether the intervention is implemented as planned.

The main questions it aims to answer is:

1. Can sufficient eligible participants be enrolled within the planned timeframe?
2. Is there any retention of participant throughout the study duration and the factors contributing to ongoing participation?
3. Can participants adhere to pre-treatment instructions and protocols before their first check-up?
4. Can participants attend and complete all assessments and chiropractic sessions?
5. Can participants fulfill all required study activities without excessive burden?
6. Can chiropractors strictly follow chiropractic adjustments only, without offering any additional treatments?

Researchers will compare adults with depression on the waitlist group to see if chiropractic care effects on adults with depression.

Participants will

* Perform resting state Electrocardiography (ECG)
* Perform resting state Electroencephalography (EEG)
* Perform Event-related potential (ERP) à Auditory and visual stimuli tests
* Complete Patient Reported Outcomes (PROs)
* COMPASS-31
* PROMIS-29
* PROMIS-Cog-8
* Perceived Stress Scale
* Depression Short Form 8a
* Complete Assessment of Acceptability
* Complete Columbia Suicide Severity Rating Scale (C-SSRS)
* Receive 6 weeks of chiropractic care treatment

DETAILED DESCRIPTION:
The investigators shall recruit 20 participants for each group, who are currently aged between 18 and 65 years and have mild to moderate depression which is measured by T score.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years of age
* Mild (T-score 55-59) to moderate (T-score 60-69) depression, as measured by the PROMIS® Depression - Short Form 8a, an 8-question survey that assesses symptoms like sadness and hopelessness.

Exclusion Criteria:

* Severe suicidal risk
* Diagnosed with any untreated or uncontrolled externalizing disorders (like substance use or antisocial disorder) or thought disorders (like schizophrenia, paranoid personality, or bipolar).
* Diagnosis of rheumatoid arthritis, osteoporosis, or cervical spine instability
* Has hearing impairments (task involves auditory stimuli)
* Currently pregnant (if applicable)
* Chiropractic adjustment within the past 2 weeks
* Scalp injuries or surgeries within the past 3 months
* Prescribed short-acting benzodiazepines, which include midazolam & triazolam
* Current litigation related to a physical, health-related injury.
* Diagnosed heart conditions, including pacemakers.
* Living with and/or caring for someone with a diagnosed neuropsychiatric disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Number of Sufficient Eligible Participants Enrolled | 1 year
  The proportion of screened participants enrolled within the recruitment timeframe. This assesses recruitment
Number of Enrolled Control Group Participants | 1 year
  Proportion of enrolled control group participants who complete the final onsite assessment. This assesses retention.
Number of Participants Who Adhere to Study | 1 year
  Proportion of enrolled participants who adhere to the pre-baseline assessment lifestyle restrictions as instructed. This assesses compliance
Number of Participants Who Chiropractic Sessions | 1 year
  Proportion of participants attending 90% of chiropractic sessions within 7 weeks. This assesses adherence to treatment
Number of Participants That Can Fulfill Study Activities | 1 year
  Proportion of participants that can fulfill all required study activities without excessive burden. This assesses tolerability

SECONDARY OUTCOMES:
Changes in Columbia Suicide Severity Scale | 1 year
  Change from baseline in suicide risk level measured using the Columbia-Suicide Severity Rating Scale (C-SSRS). This tool assesses the presence and severity of suicidal ideation and behavior using six standardized yes/no items. The outcome is the highest level of suicide risk endorsed. Higher scores indicate greater suicide risk.
Changes in COMPASS-31 | 1 year
  Changes from baseline of self-reported outcomes of neurodegenerative system symptoms utilizing the Composite Autonomic Symptom Score-3 scale. Score range from 0-100. A higher score would indicate worse autonomic symptom severity.
Changes in PROMIS-29 | 1 year
  Changes from baseline of self-reported outcomes of a comprehensive overview of a patient's physical, mental, and social health utilizing the PROMIS-29 scale. T scores range from 20-80 with a higher score indicating better health.
Changes in Perceived Stress Scale (PSS) | 1 year
  Change from baseline of self-reported symptoms of stress utilizing the Perceived Stress Scale 10. Score ranges from 0-40. A lower score indicates less stress, and a higher score indicates high stress.
Changes in PROMIS-Cog 8 | 1 year
  Changes from baseline of self-reported cognitive abilities, such as memory, attention, and decision-making utilizing the PROMIS-Cog 8 scale. T scores range from 20-80. A higher T score range indicates better cognitive functioning.
Heart Activity (ECG/HRV) | 1 year
  Change from bassline in differences in heart rate variability (HRV)
Brain Activity (Resting EEG) | 1 year
  Changes in baseline of resting-state brain wave patterns (alpha, beta, theta, delta, gamma).
Event-Related Potentials (ERP) | 1 year
  Changes from bassline in brain responses to auditory oddball stimuli (e.g., P300 and MMN components), visual oddball stimuli (e.g., N100, N200, P300 ERP components), load-picture stimuli (e.g., N100, N200, P300 ERP components) using EEG.
Change in Brain-Heart Interplay | 1 year
  Changes in baseline of brain and heart activity to understand potential mechanisms of change utilizing EEG and HRV test such as postural challenge and EEG brain wave recordings.
Assessment of Acceptability | 1 year
  Participant ratings of acceptability from the participant's perspective, including their experiences with care, interaction with providers, and overall satisfaction with study participation.
Change in PROMIS Depression 8a | 1 year
  Change from baseline in depressive symptoms measured using the PROMIS Depression Short Form 8a. This questionnaire assesses negative mood, sadness, loss of interest, hopelessness, and related depressive symptoms over the past 7 days. Raw scores from the 8 items are converted into a single PROMIS T-score 20-80, representing overall depression severity.
  Higher T-scores indicate greater depressive symptom severity.

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Chiropractic Research, Marietta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No